CLINICAL TRIAL: NCT06258772
Title: Effectiveness of Mepolizumab in the Treatment of Patients With Severe Uncontrolled CRSwNP: a Multicentric Real Life Observational Study
Brief Title: Mepolizumab in the Treatment of Patients With Severe Uncontrolled CRSwNP: a Multicentric Real Life Observational Study
Acronym: MEPOREAL
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, DE CORSO EUGENIO, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6231
Record Dates: First submitted 2024-02-02; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
MeSH Terms: interventions — mepolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Severe, uncontrolled CRSwNP patients in therapy with Mepolizumab
  Interventions: Drug: Mepolizumab Auto-Injector

INTERVENTIONS:
Drug: Mepolizumab Auto-Injector — Mepolizumab 100 mg in pre-filled injector
  Other Names: Mepolizumab 100 mg

SUMMARY:
Chronic rhinosinusitis with nasal polyposis (CRSwNP) is a complex chronic inflammatory disease of the nasosinusal mucosa that has a significant negative impact on patients' quality of life.

In CRSwNP, chronic inflammation is primarily driven by type 2 pro-inflammatory interleukins (ILs )such as IL-5, IL-4, and IL-13 along- side high levels of eosinophils in the surrounding tissue. Mepolizumab is a targeted, humanized anti-IL-5 antibody that prevents IL-5 from binding to its receptor on eosinophils and selectively inhibits eosinophilic inflammation.

So far, randomized clinical trials have assessed efficacy and safety of Mepolizumab in a large number of patients, whereas evidences in real life clinical practice are limited to few monocentric series.

Herewith, we present a multicenter, observational, prospective/retrospective nationwide real-life study with the aim to confirm the effectiveness and the safety of Mepolizumab over the first year of treatment in a real life setting.

The primary objective of this study is to evaluate the reduction of dimension of nasal polyps and the improvement of quality of life in the patient measured through symptomatologic questionnaires.

The secondary objective is to evaluate improvements in terms of smell dysfunction, comorbidities, biomarkers (nasal cytology and blood eosinophilia), need of surgery or systemic steroids.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who can sign a written informed consent Confirmed clinical / radiological diagnosis of chronic rhinosinusitis with diffuse naso-sinusal polyposis by nasal endoscopy and/or massive facial CT scan without contrast medium carried out within 6 months prior to the start of therapy;
* Blood eosinophils >150
* Severe disease stage, defined by Nasal Polyp Score (NPS) ≥ 5 or nasal obstruction symptom visual analogue scale (VAS) score of >5 and/or Sinonasal outcome tests-22 (SNOT-22) ≥ 50);
* Inadequate symptom control with intranasal local corticosteroid therapy;
* Failure of previous medical treatments (at least 2 cycles in the last year of systemic corticosteroid) and failure of previous surgical treatment through nasal endoscopic surgery (FESS), with no clinical benefit or postoperative complications.

Exclusion Criteria:

* Age <18 years;
* Patients undergoing immunosuppressive therapies;
* Patients undergoing radio/chemotherapy treatments for cancer in the 12 months before the start of therapy;
* Patients on concomitant long-term corticosteroid therapy for chronic autoimmune disorders.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We included all patients that were referred to Mepolizumab therapy, prescribed accordingly to the plan provided by AIFA
Sampling Method: Non-Probability Sample
Enrollment: 199 (Estimated)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Nasal Polyp Score | 24 months
  Evaluation of polyps volume from 0 (minimum) to 4 (maximum) points for each nasal cavity. Reduced score indicates improvement
Sinonasal Outcome Test - 22 | 24 months
  Questionnaire measuring health-related quality of life. The score is from 0 (minimum) to 110 (maximum). Reduced score indicates improvement

SECONDARY OUTCOMES:
Visual Analogue Scale for nasal obstruction | 24 moths
  Evaluation of nasal obstruction from 0 (minimum) to 10 (maximum) ;reduced score indicates improvement
Nasal Congestion Score (NCS); score (range 0-3); | 24 months
  Evaluation of nasal congestion educed score indicates improvement
Visual Analogue Scale for smell | 24 months
  Evaluation of olfaction impairment from 0 (minimum) to 10 (maximum); reduced score indicates improvement
Sniffing sticks identification test | 24 months
  Test of nasal chemosensory performance based on pen-like odor dispensing devices. From 0 (minimum ) to 16 (maximum); increased score indicates improvement.
Change in blood eosinophil count | 24 months
  Change in blood eosinophil count in a complete blood count (CBC)
Adherence to drug therapy with Mepolizumab | 24 months
  Number of missing injection in a year
Need for rescue oral corticosteroids | 24 months
  Number of oral corticosteroids cycles during therapy
Need for surgery | 24 months
  Number of surgeries performed during therapy

CONTACTS AND LOCATIONS:
Locations (27):
- Italy (27):
  - Ospedali PO di Venere e San Paolo, Bari
  - Policlinico Universitario di Bari, Ospedale Giovanni XXIII,, Bari
  - AUSL Bologna, Bologna
  - ASST degli spedali civili di Brescia,, Brescia
  - Azienda Ospedaliero Universitaria Policlinico - S. Marco,, Catania
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino,, Genova
  - Ospedale Vito Fazzi, ASL Lecce, Lecce
  - ASST Santi Paolo e Carlo, Milan
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliero-Universitaria di Modena - Modena, Modena
  - Azienda ospedaliera policlinico Federico II di Napoli, Napoli
  - Ospedale Maggiore della Carità di Novara,, Novara
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga,, Orbassano (TO)
  - Azienda Ospedaliera Università di Padova, Padua
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - Azienda Ospedaliero-Universitaria Pisana - Pisa, Pisa
  - Azienda USL - IRCCS di Reggio Emilia, Reggio Emilia
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - Fondazione Policlinico Universitario A.Gemelli IRCCS, Roma
  - Ospedaliero- Universitaria Policlinico Umberto I, Roma
  - Policlinico Tor Vergata: Fondazione PTV, Roma
  - Presidio Ospedaliero San Filippo Neri,, Roma
  - Azienda Ospedaliero- Universitaria Senese, Siena
  - i ASL ROMA 5 - Distretto Sanitario di Tivoli, Tivoli
  - ASST sette laghi Varese,, Varese

IPD SHARING:
Plan to Share IPD: Undecided